CLINICAL TRIAL: NCT04031599
Title: An Open-label, Randomized, Crossover Trial to Assess the Efficacy of Single-hormone Closed-loop System With a Rapid Acting Insulin Analogue Combined With Either Conventional Carbohydrate Counting or a Simplified Qualitative Meal-size Estimation in Regulating Glucose Levels in Adults With Type 1 Diabetes
Brief Title: Assessment of the Efficacy of the Artificial Pancreas Combined With a Qualitative Meal Size Estimation to Control Postprandial Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS18
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Artificial pancreas; Closed-loop system; Insulin; Postprandial glucose; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Motor Activity | interventions — Insulin Infusion Systems; Continuous Glucose Monitoring; Insulin Aspart; Insulin Lispro; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate counting (Active Comparator): Rapid acting insulin analogue with carbohydrate counting
  Interventions: Device: Single-hormone closed-loop system; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Aspart or Lispro; Other: Carbohydrate counting; Other: 3-week intervention; Other: 1-hour postprandial exercise (sub-study); Other: 2-hour postprandial exercise (sub-study); Other: Exercise announcement and meal bolus reduction (sub-study)
- Simplified qualitative meal size estimation (Active Comparator): Rapid acting insulin analogue with simplified qualitative meal size estimation
  Interventions: Device: Single-hormone closed-loop system; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Aspart or Lispro; Other: Simplified qualitative meal-size estimation strategy; Other: 3-week intervention

INTERVENTIONS:
Device: Single-hormone closed-loop system — Every 10 minutes, the glucose levels as measured by the sensor will be transferred automatically to a LG Google Nexus Smartphone that the algorithm is running on, which will calculate the recommended doses and will send them wirelessly to the infusion pump.
Device: Insulin pump — Tandem Diabetes Care
Device: Continuous glucose monitoring system — Dexcom G6
Drug: Aspart or Lispro — Aspart or lispro will be infused with the infusion pump
Other: Carbohydrate counting — Participants will be required to enter an estimate of the carbohydrate content of their meal into the phone. Insulin boluses will be calculated based on grams of carbohydrates and participant's insulin-to-carbohydrate ratio. Carbohydrate-matching full prandial bolus will be given 5 to 10 minutes before the meal.
  Arms: Carbohydrate counting
Other: Simplified qualitative meal-size estimation strategy — A pre-meal partial prandial bolus will be given 5-10 minutes before the meal. The partial bolus will be based on the estimated meal size (small, regular, large and extra-large). The closed-loop system will give the remaining insulin needed based on the sensor readings. For this strategy, meal size will be defined as: small as any meal less than 30g, regular meal as any meal between 30g and 60g CHO, large meal as any meal between 60g and 90g CHO, extra-large meal for anything above 90g CHO.
  Arms: Simplified qualitative meal size estimation
Other: 3-week intervention — Glucose levels will be regulated by the single-hormone closed-loop system for 3 consecutive weeks.
Other: 1-hour postprandial exercise (sub-study) — 60 minute exercise will be started one hour after the meal time.
  Arms: Carbohydrate counting
Other: 2-hour postprandial exercise (sub-study) — 60 minute exercise will be started two hours after meal time
  Arms: Carbohydrate counting
Other: Exercise announcement and meal bolus reduction (sub-study) — Meal bolus reduction of 33% at meal time and exercise announcement (increased target glucose from 6 to 9mmolL) to the CLS algorithm
  Arms: Carbohydrate counting

SUMMARY:
Postprandial glycemic excursions are major determinants of overall glycemic control in type 1 diabetes. Carbohydrate content of ingested meals is the main determinant of post-meal glucose excursion. Accurate carbohydrate counting is a critical aspect of managing postprandial blood glucose levels. accurate carbohydrate counting is considered by patients as a significant burden and frustrating task.

The closed-loop system (CLS) is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings.

The objective of this study is to compare the efficacy of two strategies to regulate glucose levels in outpatient settings in adults with type 1 diabetes: 1) single-hormone CLS with rapid acting insulin analogue combined with carbohydrate counting; 2) single-hormone CLS with rapid acting insulin analogue combined with simplified qualitative meal-size estimation.

A sub-study will also be proposed to participants. Postprandial exercise combines two situations complicating CLS operation: a high plasma insulin due to insulin on-board related to meal boluses and rapid blood glucose changes (postprandial blood glucose excursion and then drop during exercise) making input from the glucose sensor less accurate. The objective of this sub-study will be to explore the safety and efficacy of the CLS using the combined strategy of pre-meal exercise announcement and meal bolus reduction of 33% when exercise is performed 1 hour compared to 2 hours post meal time.

ELIGIBILITY:
Inclusion criteria

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. Currently using, or willing to switch to Lispro U100 or Aspart for the duration of the study.
5. HbA1c < 10%.

Exclusion criteria

1. Clinically significant nephropathy, neuropathy (e.g. known or suspected gastroparesis) or retinopathy (e.g. proliferative retinopathy) as judged by the investigator
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery
3. Anticipated need to use acetaminophen during interventions with the closed-loop system
4. Pregnancy (ongoing or current attempt to become pregnant)
5. Breastfeeding
6. No nearby third party for assistance if needed (e.g. severe hypoglycemia glucagon treatment)
7. Plans to go abroad or travel at more than 3 hours distance from Montreal during the trial period
8. Severe hypoglycemic episode within two weeks of screening or during the run-in period
9. Severe hyperglycemic episode requiring hospitalization in the last 3 months
10. Current use of glucocorticoid medication (except low stable dose and inhaled steroids)
11. Agents affecting gastric emptying (Motilium®, Victoza®, Ozempic®, Trulicity®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, Prandase®, DPP-4 inhibitors) if not at a stable dose for 3 months. Otherwise, these medications are acceptable and will be kept stable during the entire protocol.
12. Current use of SGLT-2 inhibitors unless at a stable dose for at least 3 months and appropriate ketone testing performed.
13. Known or suspected allergy to the trial products
14. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator
15. Anticipation of a significant change in exercise regimen between admission and end of the trial (i.e. starting or stopping an organized sport)
16. In the opinion of the investigator, a participant who in unable or unwilling to observed the contraindications of the study devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 10.0 mmol/L | 504 hours
Relative decrease in glucose levels during exercise compared to pre-breakfast levels (sub-study) | 3.5 or 4.5 hours
  Difference between pre-breakfast levels and the lowest glucose level from the start of the exercise until the end of exercise

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 7.8 mmol/L | 504 hours
Percentage of time of glucose levels spent below 3.9 mmol/L | 504 hours
Percentage of time of glucose levels spent below 3.3 mmol/L | 504 hours
Percentage of time of glucose levels spent below 2.8 mmol/L | 504 hours
Percentage of time of glucose levels spent above 10.0 mmol/L | 504 hours
Percentage of time of glucose levels spent above 13.9 mmol/L | 504 hours
Percentage of time of glucose levels spent above 16.7 mmol/L | 504 hours
Mean glucose levels | 504 hours
Fasting glucose levels | 504 hours
Standard deviation of glucose levels | 504 hours
Standard deviation of insulin delivery | 504 hours
Coefficient of variance of glucose levels | 504 hours
Coefficient of variance of insulin delivery | 504 hours
Between-day variability in glucose levels | 504 hours
Between-day variability in insulin delivery | 504 hours
Total insulin delivery | 504 hours
Number of hypoglycemic events less than 3.1 mmol/L | 504 hours
Number of nights with hypoglycemic events less than 3.1 mmol/L | 126 hours
Number of days with hypoglycemic events less than 3.1 mmol/L | 252 hours
Total number of hours of sensor availability | 378 hours
Percentage of time of sensor availability | 504 hours
2-hour postprandial glucose levels over the last 3 days of the intervention. | 18 hours
Average number of days per participant requiring study team support for at least one technical problem | 21 days
Number of hours and percentage of time in open-loop and closed-loop modes | 504 hours
Average number of phone calls per participant related to CLS technical issues | 504 hours
Decrease in plasma glucose levels during exercise (sub-study) | 1 hour
  Difference between glucose levels at the beginning of the exercise and the lowest glucose levels from the start of the exercise until the end of exercise
Relative decrease in glucose levels during exercise compared to pre-breakfast levels (sub-study) | 2 or 3 hours
  Difference between pre-breakfast levels and the lowest glucose level from the start of the exercise until the end of exercise
Percentage of time of plasma glucose levels spent below 3.9 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent below 3.3 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent below 3.0 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent between 3.9 and 10.0 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent above 10.0 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent above 13.9 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent above 16.7 mmol/L (sub-study) | 1 or 2 hours
  Pre-exercise period (from mealtime to exercise onset)
Percentage of time of plasma glucose levels spent below 3.9 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent below 3.3 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent below 3.0 mmol/L (sub-study) | 1 hour
  Exercise period
Number of patients experiencing hypoglycemia requiring treatment (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent between 3.9 and 10.0 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent above 10.0 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent above 13.3 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent above 16.7 mmol/L (sub-study) | 1 hour
  Exercise period
Percentage of time of plasma glucose levels spent below 3.9 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent below 3.3 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent below 3.0 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent between 3.9 and 10.0 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent above 10.0 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent above 13.3 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Percentage of time of plasma glucose levels spent above 16.7 mmol/L (sub-study) | 1.5 hour
  Post-exercise period
Number of patients experiencing hypoglycemia requiring treatment (sub-study) | 3.5 or 4.5 hours
  Overall study period
Mean time (minutes) to the first hypoglycemic event (sub-study) | 1 hour
  Exercise period

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Montreal Clinical Research Institute
Locations (2):
- Canada (2):
  - Montreal Clinical Research Institute, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Derived] Myette-Cote E, Molveau J, Wu Z, Raffray M, Devaux M, Tagougui S, Rabasa-Lhoret R. A Randomized Crossover Pilot Study Evaluating Glucose Control During Exercise Initiated 1 or 2 h After a Meal in Adults with Type 1 Diabetes Treated with an Automated Insulin Delivery System. Diabetes Technol Ther. 2023 Feb;25(2):122-130. doi: 10.1089/dia.2022.0338. Epub 2022 Dec 6. PMID 36399114